CLINICAL TRIAL: NCT06964737
Title: A Phase I, Dose-Escalation Trial of Anti-GARP Chimeric Antigen Receptor-T Cell Therapy in Patients With Recurrent High-Grade Glioma Treated at a Single Medical Center
Brief Title: Anti-GARP Chimeric Antigen Receptor T Cell Therapy for the Treatment of Recurrent Grade III or IV Gliomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, James Elder, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-24179; NCI-2025-03042 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Malignant Glioma; Recurrent WHO Grade 3 Glioma; Recurrent WHO Grade 4 Glioma; WHO Grade 2 Glioma; WHO Grade 3 Glioma; WHO Grade 4 Glioma
MeSH Terms: conditions — Glioma | interventions — Specimen Handling; X-Rays; Magnetic Resonance Spectroscopy; Blood Component Removal; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (anti-GARP CAR T cell) (Experimental): Patients undergo apheresis on day -14 and undergo surgery and placement of CSF reservoir on day 0. Patients receive anti-GARP CAR T intracavitary infusion on day 14, 21, 28, 35 and 42 in the absence of disease progression or unacceptable toxicities. Additionally, patients undergo ECHO or MUGA at screening and collection of CSF and blood samples, lumbar puncture, chest x-ray and MRI throughout the study.
  Interventions: Biological: Anti-GARP Chimeric Antigen Receptor-T Cells; Procedure: Biospecimen Collection; Procedure: Chest Radiography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Procedure: Pheresis; Procedure: Surgical Procedure

INTERVENTIONS:
Biological: Anti-GARP Chimeric Antigen Receptor-T Cells — Given intracavitary
  Other Names: Anti-GARP CAR T Cells (SY); Anti-GARP CAR T-cells (SY); Anti-GARP CAR-T Cells (SY)
Procedure: Biospecimen Collection — Undergo collection of CSF and blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Chest Radiography — Undergo chest x-ray
  Other Names: Chest X-ray
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Pheresis — Undergo apheresis
  Other Names: Apheresed; Apheresis; Blood Component Removal; Collection, Apheresis/Leukapheresis; Hemapheresis
Procedure: Surgical Procedure — Undergo surgery and placement of CSF reservoir
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of anti-glycoprotein-A repetitions predominant (GARP) chimeric antigen receptor (CAR) T cell therapy and how well it works in treating patients with grade III or IV gliomas that have come back after a period of improvement (recurrent). CAR T-cell therapy is a type of treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory so they will attack tumor cells. T cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein, such as GARP, on the patient's tumor cells is added to the T cells in the laboratory. The special receptor is called a CAR. Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain tumors. Giving anti-GARP CAR T cell therapy may be safe, tolerable, and/or effective in treating patients with recurrent grade III or IV gliomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety and feasibility of a CAR T targeting GARP for glioma by defining rate, frequency, and severity of dose limiting toxicities (DLT) following intracavity administration to patients with recurrent glioma, to determine recommended phase II dose (RP2D).

SECONDARY OBJECTIVES:

I. To describe the adverse event profile of anti-GARP CAR T cell therapy. II. To describe the cytokine levels and immunophenotype in cerebrospinal fluid (CSF) during and following anti-GARP CAR T cell therapy.

III. To describe the duration of anti-GARP CAR T cell persistence and phenotype in CSF.

IV. To describe anti-tumor activity of anti-GARP CAR T cell therapy based on objective response rate (ORR), as measured by established radiological criteria.

V. To estimate the progression-free survival (PFS) and overall survival (OS) of patients receiving anti-GARP CAR T cell therapy.

VI. For research participants with tumor specimens from primary resections and/or autopsy, describe GARP expression levels pre- and post-treatment and correlate with outcomes.

VII. To describe the frequency and phenotype of anti-GARP CAR T cells and describe GARP expression in resected post-treatment tumor tissue at progression (for patients in whom surgical resection is indicated).

EXPLORATORY OBJECTIVES:

I. To assess peripheral blood (mononuclear cells, plasma) and CSF for biomarkers that may be associated with response to anti-GARP CAR T cell therapy.

II. To assess archival tissues (primary resection), recurrent tumor, and/or autopsy specimens for biomarkers that may be associated with response to anti-GARP CAR T cell therapy.

III. To assess baseline genetic markers that may be associated with response to anti-GARP CAR T cell therapy.

OTHER EFFICACY OBJECTIVES:

I. Best overall response, determined via response assessment in neuro-oncology (RANO) criteria.

II. Clinical benefit rate that includes all subjects receiving 5 doses of anti-GARP CAR T cell therapy who demonstrate a complete response (CR), partial response (PR), or stable disease (SD) of at least 6 months duration.

III. Duration of response, calculated as the time from which a response is first observed (CR or PR) until progression or death, whichever occurs first.

IV. Overall survival (OS), calculated from first administration of study drug until death for up to two years after receiving the drug.

OUTLINE: This is a dose-escalation study.

Patients undergo apheresis on day -14 and undergo surgery and placement of CSF reservoir on day 0. Patients receive anti-GARP CAR T intracavitary infusion on day 14, 21, 28, 35 and 42 in the absence of disease progression or unacceptable toxicities. Additionally, patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) at screening and collection of CSF and blood samples, lumbar puncture, chest x-ray and magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed up at 2 weeks then at 3, 4, 6, 8, 12 and 24 months then annually for at least 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients are ≥ 18 years old
* Capacity to understand and willingness to provide written informed consent
* Diagnosis or clinical suspicion of recurrent malignant glioma, including:

  * History of high-grade glioma (World Health Organization [WHO] grade III or IV), or
  * Prior, histologically-confirmed diagnosis of grade II glioma with new radiographic findings consistent with a high-grade glioma
* Imaging and/or histopathological confirmation of recurrent disease, or verification of "high risk" histology confirmed by a biopsy with measurable disease by the Radiologic Assessment in Neuro-Oncology (RANO) criteria
* Disease in one hemisphere and is supratentorial
* If on steroids such as dexamethasone, must be on a low dose (≤ 4mg per day) at the time of treatment, and not at an ascending dosage schedule at time of enrollment/leukapheresis
* Subjects must not have received bevacizumab therapy and are not planned to start such therapy
* Karnofsky performance score (KPS) ≥ 60
* Surgical candidate for surgery for malignant glioma
* White blood cells (WBC) > 4,000 cells/uL
* Hemoglobin (Hgb) > 7 gm/dL
* Platelets (Plt) > 100/dL
* Serum creatinine ≤ 1.5 x institutional upper limit of normal
* Liver function tests within 1.5 x institutional upper limit of normal
* Women of reproductive potential must have a negative pregnancy test within 7 days of study start. All patients of reproductive potential must use a physician-approved contraceptive and refrain from sperm donation for at least two weeks prior, during, and six months after final T cell infusion. Women must refrain from breastfeeding for six months after final T cell infusion
* Sufficient venous access, to be confirmed prior to apheresis

Exclusion Criteria:

* Patients who have a history of malignancy other than the glioma under investigation in this study, except patients with the following malignancies/treatment characteristics, who are eligible at the investigator's discretion:

  * Patients with a history of malignancy that has been treated with curative intent at least 2 years prior to screening and with no evidence of relapse, if no concurrent anti-cancer therapy (except hormonal therapy) is being given
  * Patients with a history of malignancy with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%) such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or stage I uterine cancer
  * Patients who have prostate cancer with no evidence of metastatic disease and are not on active therapy, except anti-androgen therapy
* History of autoimmune disease, or other diseases require long-term administration of high-dose steroids [> 10 mgs/day] or immunosuppressive therapies

  * Research participants who received steroids must have either received their last dose of steroids 7 days or more prior to apheresis or have dosage tapered to < 2mg/kg/day
* Patients being treated concurrently (within 14 days prior to study enrollment) with any other investigational agent

  * Examples of other investigational agents that would be exclusionary include supportive care agents
* Patients receiving anti-cancer agents such as chemotherapy (e.g., temozolomide) must stop treatment 14 days prior to undergoing apheresis and remain off therapy throughout the duration of CAR T therapeutic intervention
* Patients with active fungal, bacterial, viral, or other infection that requires intravenous antimicrobials

  * Prophylactic antimicrobials are allowed
  * Patients with active invasive fungal infection should be excluded even if the treatment is oral antimicrobials
* History of allergy to study products/diluents/emulsions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities | Up to 30 days after the first dose
  The rate, frequency and severity will be defined using Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5. Will be summarized by descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days after last dose of study drug
  The rate, frequency and severity will be defined using CTCAE v 5. Will be summarized by descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Cytokine levels and immunophenotype in cerebrospinal fluid (CSF) | During and following therapy, assessed up to 15 years
Duration of anti-glycoprotein-A repetitions predominant (GARP) chimeric antigen receptor (CAR) T cell persistence and phenotype in CSF | Up to 15 years
Objective response rate (ORR) | Up to 15 years
  ORR will be calculated and exact binomial 95% confidence interval (CI) will be provided.
Progression-free survival (PFS) | From initiation of therapy to the time of progression or death, assessed up to 15 years
  Kaplan-Meier methods will be used to estimate PFS with 95% CI.
Overall survival (OS) | From initiation of therapy to death, assessed up to 15 years
  Kaplan-Meier methods will be used to estimate OS with 95% CI.
Correlation of GARP expression levels with outcomes | At pre- and post-treatment, assessed up to 24 months
  Relative GARP expression in tumor tissue will be summarized using descriptive statistics.
Frequency and phenotype of anti-GARP CAR T cells in tumor tissue | At progression, assessed up to 15 years
  The level and phenotype of anti-GARP CAR T in tumor tissue will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: James B Elder, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Wu BX, Kreatsoulas D, Cam H, Bolyard C, Chang Y, Mandula J, Welsh PW, Wang Z, Li A, Weltge P, Elder JB, Giglio P, Otero JJ, Rajappa P, Gerald D, Chung D, Ma Q, Velegraki M, Li Z. Targeting TGFbeta docking receptor Glycoprotein A Repetitions Predominant (GARP) via novel chimeric antigen receptor (CAR)-T cell platform to treat glioblastoma. Neuro Oncol. 2025 Aug 27:noaf195. doi: 10.1093/neuonc/noaf195. Online ahead of print. PMID 40873341
- See also: The Jamesline — http://cancer.osu.edu